CLINICAL TRIAL: NCT01815606
Title: Randomized Trial Comparing 19 and 25G Needles for Fine Needle Aspiration (FNA) of Solid Pancreatic Mass Lesions Greater Than 35mm
Brief Title: Trial Comparing 19 and 25G Needles for Fine Needle Aspiration (FNA) of Solid Pancreatic Mass Lesions Greater Than 35mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 405581
Record Dates: First submitted 2013-02-26; First posted 2013-03-21 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; cancer; EUS-FNA; 19Gauge; 25Gauge; 35mm mass
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 19 Gauge needle biopsy (Active Comparator): biopsy with 19 gauge needle
  Interventions: Procedure: biopsy with 19 gauge needle
- 25 gauge needle biopsy (Active Comparator): biopsy with 25 gauge needle
  Interventions: Procedure: biopsy with 25 gauge needle

INTERVENTIONS:
Procedure: biopsy with 19 gauge needle — biopsy with 19 gauge needle
  Other Names: FNA; biopsy
  Arms: 19 Gauge needle biopsy
Procedure: biopsy with 25 gauge needle — biopsy with 25 gauge needle
  Other Names: FNA; biopsy
  Arms: 25 gauge needle biopsy

SUMMARY:
This study will test two different needles for performing a biopsy of the pancreas during endoscopic ultrasound (EUS) procedures. Patients who are asked to participate in this study have a growth in the pancreas measuring greater than 35mm that needs a biopsy so that a diagnosis can be made. The biopsy can be performed using either a 19 or 25-Gauge needle. The purpose of this study is to compare which of the two needles is better for performing biopsies of the pancreas on masses that are greater than 35mm.

DETAILED DESCRIPTION:
Endoscopic Ultrasound-guided fine needle aspiration (EUS-FNA) can be performed using the 25, 22 or 19 gauge (G) needles. Randomized trials have shown that all three needles are safe and perform equally well. However, in a retrospective study, the diagnostic sensitivity of EUS-FNA for pancreatic masses that measured more than 35mm was less compared to smaller size masses. This is because larger size tumors have more necrosis and it is difficult to identify cancer cells in them to make a diagnosis. Therefore, more biopsies must be performed in larger size tumors to establish a diagnosis. In previous studies it has been shown that the larger 19G needles procure larger and better quality tissue. Therefore, our hypothesis is that, when a larger 19G needle is used to FNA tumors more than 35mm, a diagnosis can be achieved with fewer passes.

ELIGIBILITY:
Inclusion Criteria:

All patients referred to Florida Hospital Endoscopy Unit for assessment of pancreatic mass lesions greater than 35 mm on computed tomography (CT) that require FNA.

Exclusion Criteria:

* Age < 19 years
* Unable to safely undergo EUS for any reason
* Coagulopathy (INR >1.6, Prothrombin Time >18secs, Thrombocytopenia <80,000 cells/ml)
* Unable to consent
* Non-English speaking patients
* Participation in any other clinical trial (excluding registries or databases)

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of passes | Up to 12 months
  The use of a 19G FNA needle reduces the number of passes required to establish a diagnosis in pancreatic tumors that are greater than 35mm in size. This translates to less sedation, faster patient recovery, better safety and time efficiency.

SECONDARY OUTCOMES:
Rate of Complication | Up to 12 months
  To compare the rate of complications associated with the 19G and 25G needles when sampling pancreatic tumors greater than 35mm in size.
  Also, the rate of needle dysfunction will be compared. Needle dysfunction is defined as, the need to use more than one needle per pancreatic tumor in an individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No